CLINICAL TRIAL: NCT01982682
Title: A Two Step Approach to Allogeneic Hematopoietic Stem Cell Transplantation for High-Risk Hematologic Malignancies Using One Haploidentical Donor
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation for High-Risk Hematologic Malignancies Using One Haploidentical Donor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13D.352; 2013-031 (Other: CCRRC); JT 2974 (Other: JeffTrial Number)
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Results first posted 2018-06-07 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic/Lymphoid Cancer
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Whole-Body Irradiation; Cyclophosphamide; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (TBI, DLI, cyclophosphamide, CD34+ donor HSCT) (Experimental): CONDITIONING REGIMEN: Patients undergo TBI BID on days -10 to -8, undergo DLI on day -6, and receive cyclophosphamide IV over 2 hours on days -3 and -2.
  TRANSPLANT: Patients undergo CD34+ (cluster of differentiation 34+) selected allogeneic HSCT on day 0.
  GVHD PROPHYLAXIS: Patients receive tacrolimus IV or PO beginning on day -1 with taper beginning by day 42, and mycophenolate mofetil IV BID on days -1 to 28.
  Interventions: Radiation: Total-Body Irradiation (TBI); Biological: Donor Lymphocyte Infusion (DLI); Drug: Cyclophosphamide; Procedure: Allogeneic hematopoietic stem cell transplantation (HSCT); Drug: Mycophenolate mofetil

INTERVENTIONS:
Radiation: Total-Body Irradiation (TBI) — Undergo TBI
Biological: Donor Lymphocyte Infusion (DLI) — Undergo DLI
Drug: Cyclophosphamide — Given IV
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune; cytophosphane; Lyophilizedcytoxan
Procedure: Allogeneic hematopoietic stem cell transplantation (HSCT) — Undergo CD34+ selected allogeneic HSCT
Drug: Mycophenolate mofetil — Given IV
  Other Names: CellCept

SUMMARY:
This phase II trial studies how well total-body irradiation, donor lymphocyte infusion, and cyclophosphamide before donor stem cell transplant works in treating patients with high-risk hematologic malignancies. Giving total-body irradiation, donor lymphocyte infusion, and chemotherapy before a donor stem cell transplant helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When certain stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Removing the T cells from the donor cells before transplant and giving tacrolimus and mycophenolate mofetil may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1) To assess 1 year relapse free survival in high risk patients undergoing hematopoietic stem cell transplant (HSCT) using the Thomas Jefferson University (TJU) 2 step approach with 2 days inserted between the last fraction of total-body irradiation (TBI) and the infusion of donor T cells (donor lymphocyte infusion [DLI]).

SECONDARY OBJECTIVES:

1. To assess regimen related toxicity in this updated conditioning regimen, graft-versus-host disease (GVHD) incidence and severity, and overall survival in patients undergoing treatment on this protocol.
2. To assess the consistency and pace of engraftment.
3. To assess the pace of T cell and B cell immune recovery.

OUTLINE:

CONDITIONING REGIMEN: Patients undergo TBI twice daily (BID) on days -10 to -8, undergo DLI on day -6, and receive cyclophosphamide intravenously (IV) over 2 hours on days -3 and -2.

TRANSPLANT: Patients undergo cluster of differentiation (CD) 34+ selected allogeneic HSCT on day 0.

GVHD PROPHYLAXIS: Patients receive tacrolimus IV or orally (PO) beginning on day -1 with taper beginning by day 42, and mycophenolate mofetil IV BID on days -1 to 28.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. This treatment is for patients with high risk hematologic malignancies. High risk is defined as:

   * Any patient with a hematologic malignancy with residual disease after treatment with 1 or more chemotherapy regimens in whom achievement of remission with additional chemoradiotherapy is felt to be unlikely
   * Patients without morphologic evidence of disease but with high risk features which would predict for relapse despite remission at HSCT such as adverse cytogenetics, 3rd or greater CR (complete response), or failure to recover peripheral blood counts to normal ranges. While these patients do not have detectable disease by current methods, like all patients they have non-detectable disease which in their case is highly aggressive.
2. Patients must have one related donor who is HLA (human leukocyte antigen) mismatched in the GVHD direction at two or more HLA loci
3. Patients must adequate organ function:

   * LVEF (left ventricular ejection fraction) of >50 %
   * Diffusing capacity of the lungs for carbon monoxide (DLCO) (adjusted for hemoglobin) >50 % of predicted and forced expiration to the full FEV-1 >50 %
   * Adequate liver function as defined by a serum bilirubin <1.8, AST (aspartate aminotransferase) or ALT (alanine aminotransferase) < 2.5X upper limit of normal
   * Creatinine clearance of > 60 ml/min
4. Karnofsky Performance Status (KPS) of > 80% on the modified (KPS) tool
5. Patients must be willing to use contraception if they have childbearing potential
6. Able to give informed consent

Exclusion Criteria:

1. Modified (KPS) Karnofsky Performance status of <80%
2. > 5 Comorbidity Points on the Hematopoietic cell transplantation - specific comorbidity (HCT-CI) Index (See Appendix B)
3. Class I or II antibodies against donor human leukocyte antigens (HLA)
4. HIV positive
5. Active involvement of the central nervous system with malignancy
6. Psychiatric disorder that would preclude patients from signing an informed consent
7. Pregnancy, or unwillingness to use contraception if they have child bearing potential
8. Patients with life expectancy of < 6 months for reasons other than their underlying hematologic/oncologic disorder
9. Alemtuzumab treatment within 8 weeks of HSCT admission
10. Anti-thymocyte globulin (ATG) level of > 2 ugm/ml
11. Patients with active inflammatory processes including T max >101 or active tissue inflammation are excluded
12. Inability to tolerate cyclophosphamide or undergo total body irradiation at the doses specified in the treatment plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-11-04 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Grosso, DNP, CRNP, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (TBI, DLI, Cyclophosphamide, CD34+ Donor HSCT): CONDITIONING REGIMEN: Patients undergo TBI BID (bis in die/ twice a day) on days -10 to -8, undergo DLI on day -6, and receive cyclophosphamide IV over 2 hours on days -3 and -2.
  TRANSPLANT: Patients undergo cluster of differentiation 34+ (CD34+) selected allogeneic HSCT on day 0.
  GVHD PROPHYLAXIS: Patients receive tacrolimus IV or PO beginning on day -1 with taper beginning by day 42, and mycophenolate mofetil IV BID on days -1 to 28.
  Total-Body Irradiation (TBI): Undergo TBI
  Donor Lymphocyte Infusion (DLI): Undergo DLI
  Cyclophosphamide: Given IV
  Allogeneic hematopoietic stem cell transplantation (HSCT): Undergo CD34+ selected allogeneic HSCT
  Mycophenolate mofetil: Given IV
Period: Overall Study
Arm/Group | Treatment (TBI, DLI, Cyclophosphamide, CD34+ Donor HSCT)
Started | 41
Completed | 40
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment (TBI, DLI, Cyclophosphamide, CD34+ Donor HSCT): CONDITIONING REGIMEN: Patients undergo TBI BID on days -10 to -8, undergo DLI on day -6, and receive cyclophosphamide IV over 2 hours on days -3 and -2.
  TRANSPLANT: Patients undergo CD34+ selected allogeneic HSCT on day 0.
  GVHD PROPHYLAXIS: Patients receive tacrolimus IV or PO beginning on day -1 with taper beginning by day 42, and mycophenolate mofetil IV BID on days -1 to 28.
  Total-Body Irradiation (TBI): Undergo TBI
  Donor Lymphocyte Infusion (DLI): Undergo DLI
  Cyclophosphamide: Given IV
  Allogeneic hematopoietic stem cell transplantation (HSCT): Undergo CD34+ selected allogeneic HSCT
  Mycophenolate mofetil: Given IV
Arm/Group | Treatment (TBI, DLI, Cyclophosphamide, CD34+ Donor HSCT)
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 24
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants That Experience 1 Year Relapse Free Survival After Undergoing Hematopoietic Stem Cell Transplantation (HSCT) Using the Thomas Jefferson University 2 Step Approach
Time Frame: Up to 1 year after HSCT
Population: One subject was inevaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (TBI, DLI, Cyclophosphamide, CD34+ Donor HSCT)
Number analyzed (Participants) | 40
Participants | 27

2. Secondary Outcome: Number of Participants With Successful Engraftment
Description: Will be reported descriptively. Successful engraftment is defined as ANC (absolute neutrophil count, the number of white blood cells (WBCs) that are neutrophils) ≥ 0.5x109/L for at least 30 days and Platelet engraftment > 20,000 with no transfusion x 7 days.
Time Frame: Up to 1 year after HSCT
Population: One subject was inevaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (TBI, DLI, Cyclophosphamide, CD34+ Donor HSCT)
Number analyzed (Participants) | 40
Participants | 37

3. Secondary Outcome: Count of Participants That Experienced Death as a Result of Graft-versus-host Disease (GVHD)
Description: Graft versus host disease was clinically characterized based on 4 stages of progression for three major body areas, skin, liver, gut. Subjects who experienced life threatening reactions in their skin, liver and gut ultimately experienced functional impairment and expired.
  Life threatening reactions in the Skin were characterized by desquamation (the shedding of the outer layers of skin) and bullae (a bubblelike cavity filled with air or fluid, in particular).
  Life threatening reactions in the Liver were characterized by Bilirubin, > 15 mg/dl Life threatening reactions in the Gut were characterized by Pain +/- ileus (a painful obstruction of the ileum or other part of the intestine.)
Time Frame: Up to 1 year after HSCT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (TBI, DLI, Cyclophosphamide, CD34+ Donor HSCT)
Number analyzed (Participants) | 40
Participants | 2

4. Secondary Outcome: Median Pace of T Cell Immune Recovery at 28 Days Post Hematopoietic Stem Cell Transplantation (HSCT)
Description: An excess amount of residual T-lymphocytes in the Peripheral Blood Stem Cell Collection (PBSC) product may increase the risk of GVHD. The ideal amount of T-cells left in the PBSC product is no greater than 5x104/kg. Every effort will be made to keep T-cell amounts to below this threshold. The median pace of T-cell immune recovery at 28 days will be monitored by collecting cluster of differentiation (CD24) and (CD38).
Time Frame: At 28 days post HSCT
Population: 3 subjects were not evaluable for this outcome measure.
Measure: Median (Full Range); unit: cells/ul
Arm/Group | Treatment (TBI, DLI, Cyclophosphamide, CD34+ Donor HSCT)
Number analyzed (Participants) | 37
cells/ul
  Median CD3/4 count at d+28 | 41.3 [9.0 to 417.0]
  Median cluster of diff. 38 (CD3/8) count at d+28 | 48 [7.9 to 1329.0]

5. Secondary Outcome: Median Pace of T Cell Immune Recovery at 90 Days Post Hematopoietic Stem Cell Transplantation (HSCT)
Description: An excess amount of residual T-lymphocytes in the Peripheral Blood Stem Cell Collection (PBSC) product may increase the risk of GVHD. The ideal amount of T-cells left in the PBSC product is no greater than 5x104/kg. Every effort will be made to keep T-cell amounts to below this threshold. The median pace of T-cell immune recovery at 90 days will be monitored by collecting cluster of differentiation (CD24) and (CD38).
Time Frame: 90 days post HSCT
Population: 5 subjects were not evaluable for this outcome measure.
Measure: Median (Full Range); unit: cells/ul
Arm/Group | Treatment (TBI, DLI, Cyclophosphamide, CD34+ Donor HSCT)
Number analyzed (Participants) | 35
cells/ul
  Median CD3/4 count at d+90 | 141 [22 to 1374]
  Median CD3/8 count at d+90 | 384 [8.4 to 3041]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment (TBI, DLI, Cyclophosphamide, CD34+ Donor HSCT)
All-Cause Mortality (participants affected / at risk) | 16/40
Serious Adverse Events (participants affected / at risk) | 32/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (TBI, DLI, Cyclophosphamide, CD34+ Donor HSCT) (N=40)
Diplopia (Eye disorders) | 1 (1)
Abdominal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (5)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Altered Mental Status (Psychiatric disorders) | 4 (4)
Blood in Stool with AVM (Gastrointestinal disorders) | 1 (1)
C. diff infection (Infections and infestations) | 1 (1)
Cardiac Disorder (Cardiac disorders) | 1 (1)
CMV reactivation (Infections and infestations) | 4 (4)
Dehydration (General disorders) | 1 (1)
Fall (General disorders) | 1 (1)
Fever (Infections and infestations) | 1 (1)
Graft rejection (General disorders) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematuria (Blood and lymphatic system disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatobiliary issue (Hepatobiliary disorders) | 1 (1)
Hyperbilirubin (Blood and lymphatic system disorders) | 6 (6)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypocellular marrow (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Vascular disorders) | 5 (5)
Hypovolemia (Blood and lymphatic system disorders) | 1 (1)
Hypoxia (Blood and lymphatic system disorders) | 11 (13)
Infection (Infections and infestations) | 4 (4)
Klesiella/enterobacteruosepsis with bacteremia (Infections and infestations) | 1 (1)
Lung Abcess (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Malaise (Gastrointestinal disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhino/enterovirus (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 4 (4)
Sleep apnea Desaturation (General disorders) | 1 (1)
Slurred Speech (General disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Syncope (Blood and lymphatic system disorders) | 1 (2)
Upper Extremity Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (TBI, DLI, Cyclophosphamide, CD34+ Donor HSCT) (N=40)
Atrial Fibrillation (Cardiac disorders) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 7 (7)
Abdominal protuberance (Musculoskeletal and connective tissue disorders) | 1 (1)
Aches (General disorders) | 2 (2)
Acid reflux (Gastrointestinal disorders) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 5 (5)
Agitated (General disorders) | 2 (2)
Altered Mental state (Psychiatric disorders) | 1 (1)
Anal fissure (Skin and subcutaneous tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Ascites (Musculoskeletal and connective tissue disorders) | 3 (3)
Asytole (Cardiac disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
BK virus (Infections and infestations) | 1 (1)
Bladder Spasm (Renal and urinary disorders) | 1 (1)
Blood in stool (Gastrointestinal disorders) | 1 (1)
Blurry vision (Eye disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 6 (6)
Chest pain (General disorders) | 4 (4)
Chest pain (infection) (Infections and infestations) | 2 (2)
Chills (General disorders) | 8 (8)
Clostridium difficile (Infections and infestations) | 3 (3)
Confusion (Psychiatric disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cranial nerve deficits (Nervous system disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 3 (3)
Cytomegalovirus (Infections and infestations) | 7 (7)
Decreased Appetite (General disorders) | 4 (4)
Decreased Ejection fraction (General disorders) | 1 (1)
Decreased intake (General disorders) | 1 (1)
Decreased Urine Output (Renal and urinary disorders) | 7 (8)
Dehydration (General disorders) | 2 (2)
Depression (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 34 (35)
Dizziness (General disorders) | 5 (5)
Double vision (Eye disorders) | 1 (1)
Dry eyes (Eye disorders) | 2 (2)
Dry Mouth (General disorders) | 6 (6)
Deep vein thrombosis (Blood and lymphatic system disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
Edema (General disorders) | 6 (6)
Electrolyte imbalance (General disorders) | 2 (2)
Elevated glucose (Hepatobiliary disorders) | 1 (1)
Emesis (Gastrointestinal disorders) | 2 (2)
Epistaxis (Blood and lymphatic system disorders) | 1 (1)
Erythemia (Skin and subcutaneous tissue disorders) | 1 (1)
Fall (General disorders) | 3 (3)
Fatigue (General disorders) | 2 (2)
Fever (Infections and infestations) | 36 (43)
Flatus (Gastrointestinal disorders) | 1 (1)
Fluid Overload (General disorders) | 12 (12)
General pain (General disorders) | 2 (2)
Hallucinations (Psychiatric disorders) | 4 (4)
Headache (General disorders) | 10 (10)
Heartburn (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 5 (5)
Hepatic Failure (Hepatobiliary disorders) | 1 (1)
HHV6 reactivation (Infections and infestations) | 5 (5)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 10 (10)
Hypertension (Blood and lymphatic system disorders) | 8 (8)
Hypokalemia (Blood and lymphatic system disorders) | 2 (2)
Hypomagnesemia (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Blood and lymphatic system disorders) | 8 (9)
Hypoxia (General disorders) | 7 (7)
Increased Creatine (Blood and lymphatic system disorders) | 3 (3)
Increased LFTs (Hepatobiliary disorders) | 3 (3)
Indigestion (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2)
infusion reaction (Product Issues) | 1 (1)
Insomnia (General disorders) | 8 (8)
Intravenous immune globulin reaction (Immune system disorders) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 4 (4)
Lethargy (General disorders) | 9 (9)
LFT abnormality (Hepatobiliary disorders) | 2 (2)
Lightheadedness (General disorders) | 1 (1)
Loose stools (Gastrointestinal disorders) | 1 (1)
Lower Extremity Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 38 (38)
Muscle pains (Musculoskeletal and connective tissue disorders) | 10 (15)
Nausea (General disorders) | 13 (13)
Neuropathy (Nervous system disorders) | 6 (6)
Neutropenic fever (Infections and infestations) | 1 (1)
Orthostasis (Blood and lymphatic system disorders) | 2 (2)
Panic attack (Psychiatric disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 6 (6)
Parotitis (Infections and infestations) | 6 (6)
Peeling skin (Skin and subcutaneous tissue disorders) | 2 (2)
Pericardial Effusion (Cardiac disorders) | 2 (2)
Pericatheter Thrombus (Blood and lymphatic system disorders) | 1 (1)
Perineal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pharyngeal edema (General disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Platelet Transfusion Reaction (General disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pruritis rash (Skin and subcutaneous tissue disorders) | 3 (3)
Pseudomonas bacteremia (Infections and infestations) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 22 (23)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Rhinoenterovirus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rigors (General disorders) | 3 (3)
Scrotal swelling (Reproductive system and breast disorders) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Sinus pain (Ear and labyrinth disorders) | 3 (3)
Skin breakdown (Skin and subcutaneous tissue disorders) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Splenomegaly (Renal and urinary disorders) | 1 (1)
Sweats (General disorders) | 1 (1)
Swelling (General disorders) | 2 (2)
Syncopal episode (Blood and lymphatic system disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 10 (11)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Thrush (Infections and infestations) | 2 (2)
Tremor (Musculoskeletal and connective tissue disorders) | 5 (5)
Trouble breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Trouble sleeping (General disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 5 (5)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Urinary Urgency (Renal and urinary disorders) | 1 (2)
UTI (Renal and urinary disorders) | 4 (4)
Ventricular tachychardia (Cardiac disorders) | 1 (1)
Visual Disturbance (Eye disorders) | 1 (1)
Volume overload (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (9)
Weakness (General disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-12-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT01982682/Prot_SAP_000.pdf
  • Informed Consent Form (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT01982682/ICF_001.pdf